CLINICAL TRIAL: NCT02174666
Title: The Effects of Red Clover Treatment on Bone Tissue Regulation in Postmenopausal Osteopenia.
Brief Title: Isoflavone Treatment for Postmenopausal Osteopenia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: European Regional Development Fund (Other); The Ministry of Science, Technology and Innovation, Denmark (Other Government)
Responsible Party: Principal Investigator, Per Bendix Jeppesen, Associate Prof., PhD, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KLKN 14-04-2014; DASTI (Other: The Ministry of Science, Technology and Innovation, Denmark)
Record Dates: First submitted 2014-06-19; First posted 2014-06-25 (Estimated); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Osteopenia; Osteoporosis
Keywords: Aglycones; Isoflavones; Red clover; Osteopenia; Menopause; Bone turnover; Bone mineral density
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis | interventions — formononetin; biochanin A; Genistein; daidzein; Vitamin D; Magnesium; Calcium; Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Red clover extract (Active Comparator): Group recieving daily red clover extract containing isoflavones (80 mg/d), along with calcium (1040 mg/d), vitamin D (25µg/d) and magnesium (487mg/d).
  Interventions: Dietary Supplement: Red clover extract
- Placebo group (Placebo Comparator): Group recieving daily placebo extract (with no isoflavone content), calcium (1040 mg/d), vitamin D (25µg/d) and magnesium (487mg/d).
  Interventions: Dietary Supplement: Supplementation (placebo)

INTERVENTIONS:
Dietary Supplement: Red clover extract — Aglycone isoflavones 80mg/d
  Other Names: Formononetin; Biochanin A; Genistein; Daidzein; Vitamin D; Magnesium; Calcium
  Arms: Red clover extract
Dietary Supplement: Supplementation (placebo)
  Other Names: Vitamin D; Magnesium; Calcuim
  Arms: Placebo group

SUMMARY:
The aim of the project is to execute a double-blind, parallel, randomized 12-month intervention trial on postmenopausal women with osteopenia (low bone mineral density), in order to determine the effects of daily intake of fermented red clover (RC) extract on estrogen dependent bone mineral resorption when compared to placebo. Both groups will recieve equivalent daily calcium, vitamin D and magnesium supplements. The project will also assess whether bioactive compounds in RC can reduce the risk of developing cardiovascular disease.

DETAILED DESCRIPTION:
The project aims to determine whether red clover derived isoflavones have capabilities to exert positive effects in conditions of osteoporosis and osteopenia in states estrogen deficiency and/or dysregulation.

The cause of osteopenia in women is thought to arise from the deficiency of and/or dysregulation by estrogen on target tissues. Hormone Replacement Therapy (HRT) has proven to be an effective treatment, however it retains limited use as there is general consensus that it also increases cancer risk. Plant derived compounds that emulate the chemical structure and behaviour of estrogen (known as isoflavones) offer a compelling alternative to HRT, due to their potential to adopt the regulatory roles of estrogen without incurring equivalent negative side effects of HRT.

There are, at present, few or no direct head to head clinical trials assessing combination treatments of isoflavones, vitamin D and calcium in contrast to standard vitamin D and calcium supplementation proscribed to osteopenic patients. Research in this area will therefore provide valuable insight into the effectiveness of isoflavones to reduce resorption and/or to stimulate the formation of bone tissue. Moreover the study will provide a comprehensive assessment of the potential of isoflavones to enhance the efficacy of existing preventative treatments. Outcomes of the project have the prospect to help thousands of middle aged and PM women suffering. Moreover, the project may enable development of functional foods and/or nutraceuticals that can be used as either a preventative measure and/or as a treatment for osteoporosis in states of estrogen deficiency and thereby provide an alternative to Hormone Replacement Therapy that does involve the same side effects and risks.

ELIGIBILITY:
Inclusion criteria:

* Age 50-85 years, only women
* Have osteopenia (T score between -1 and -2.5)
* Body Mass Index (BMI) between 20 and 40

Exclusion criteria:

* Taken specific osteoporosis drugs (i.e. bisphosphonates, PTH, estrogen or strontium ranelate) in the past 3 months
* Taken other selective estrogen receptor modulator preparations (raloxifene, tamoxifen or isoflavones) in the past 3 months
* Participation in other clinical trials within the last 3 months
* Previous history of cardiovascular, psychiatric, neurological, and / or kidney disease
* Alcohol or substance abuse or acute illness
* Blood pressure> 160/110
* Pregnant and breastfeeding women

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Plasma C-terminal telopeptide (CTX) | 0 - 12 months
  Bone mineral resorption biomarker.

SECONDARY OUTCOMES:
Bone mineral density via dual energy X-ray absorptiometry | 0 - 12 months
  Objective measure of bone mineral density and bone mineral content.

CONTACTS AND LOCATIONS:
Overall Officials: Per B Jeppesen, Prof PhD, Principal Investigator — Department of Medicine and Endocrinology MEA, Aarhus University
Locations (1):
- Aarhus University Hospital, Aarhus, Central Jutland, Denmark

REFERENCES:
- [Derived] Lambert MNT, Thybo CB, Lykkeboe S, Rasmussen LM, Frette X, Christensen LP, Jeppesen PB. Combined bioavailable isoflavones and probiotics improve bone status and estrogen metabolism in postmenopausal osteopenic women: a randomized controlled trial. Am J Clin Nutr. 2017 Sep;106(3):909-920. doi: 10.3945/ajcn.117.153353. Epub 2017 Aug 2. PMID 28768651